CLINICAL TRIAL: NCT06158646
Title: Mechanically or Kinematically Aligned Total Knee Prosthesis: Prospective and Comparative Study of Clinical, Stereoradiographic, and Biomechanical Results
Brief Title: Mechanically or Kinematically Aligned Total Knee Prosthesis
Acronym: BIOMAKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Sport, Bordeaux Mérignac (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01312-43
Record Dates: First submitted 2023-11-14; First posted 2023-12-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Knee
Keywords: total knee prosthesis; mechanical alignment; kinematic alignment; biomechanic study
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with kinematic aligned knee prosthesis (Experimental)
  Interventions: Device: kinematic knee prosthesis
- patients with biomechanic aligned knee prosthesis (Active Comparator)
  Interventions: Device: biomechanic knee prosthesis

INTERVENTIONS:
Device: kinematic knee prosthesis — Patients with a kinematically aligned total knee prosthesis and having a post-operative follow-up consultation within at least 1 year after their surgery are consecutively pre-selected according to the eligibility criteria.
  Arms: patients with kinematic aligned knee prosthesis
Device: biomechanic knee prosthesis — A group of patients with a mechanically aligned TKA and scheduled for a follow-up consultation 1 year after surgery will be identified to be matched on the aforementioned criteria (sex, age, BMI).
  Arms: patients with biomechanic aligned knee prosthesis

SUMMARY:
The mechanical alignment technique (Mechanical Alignment - MA) of a total knee prosthesis (TKA) was developed with the aim of making the installation of a TKA simple and reproducible, and that the prosthetic biomechanics are acceptable, thus promoting good longevity of implants. This is a technique that does not aim to restore the constitutional anatomy of the knee; bone cuts are systematically made at fixed angles, in the 3 planes of space, in relation to the mechanical axes of the long bones (femur and tibia). This non-personalized implantation technique therefore systematically alters the anatomy, laxity and kinematics of the knee, causing up to 50% of residual symptoms after prosthetic implantation and 20% of dissatisfied patients.

In order to improve the clinical results of TKA, a new, more personalized and physiological technique was developed in 2007, called Kinematic Alignment (KA). This technique aims to restore the pre-arthritic anatomy, unique to each knee. Patients with severe constitutional deformity of the lower limb therefore retain this deformity after kinematic prosthetic replacement. The impact of the alignment technique on the biomechanics of the prosthetic knee remains poorly described. The main objective of this study is therefore to compare knee biomechanics between mechanical TKA and kinematic TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed as part of a consultation 1 year after TKA placement
* Adult patient
* Patient affiliated to a social security system
* Patient informed of the study and formally included (signing of informed consent) before the first research review

Exclusion Criteria:

* Patient with a contralateral knee prosthesis
* Patient with another condition (acquired pathology) of the lower limbs (e.g. severe osteoarthritis of the contralateral knee or hip/ankle) and/or of the nervous system (e.g. Parkinson's) which may significantly affect the quality of walking
* Pregnant patient
* Patient deprived of liberty by judicial or administrative decision,
* Adult patient subject to a legal protection measure or unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Biomechanical parameters of knee : spatiotemporal parameters | One year after surgery
  When walking on flat ground and when going up/down stairs:
  walking speed
Biomechanical parameters of knee : Kinematic parameters in the 3 planes of space | One year after surgery
  dynamic hip-knee-ankle angles during the knee flexion/extension test with and without support
Biomechanical parameters of knee : joint moments | One year after surgery
  Unit : Newton meter
Biomechanical parameters of knee : force | One year after surgery
  Unit : body weight
Biomechanical parameters of knee : lever arms | One year after surgery
Symmetry index between the operated limb and the healthy controlateral limb | One year after surgery
  Comparison between the two limbs

SECONDARY OUTCOMES:
Clinical results : Patient-Reported Outcome Measures: Functional score (OXFORD scale) | One year after surgery
  OXFORD scale : numerical rating scale used to quantify the power or strength produced by the contraction of a muscle (0-5) ; 5 is maximal strenght
Clinical results : Patient-Reported Outcome Measures: joint perception score | One year after surgery
  Forgotten joint score : joint-specific questionnaire that focuses on the patients' awareness of their prosthetic joint during daily activities ; 0-100 (0 is the worst result and 100 the better result possible)
Clinical results : Patient-Reported Outcome Measures: pain | One year after surgery
  visual analog scale (VAS) pain (numerical scale 0-10), 0 is absence of pain and 10 the worst pain possible
Clinical results : Patient satisfaction | One year after surgery
  Scale from "not at all satisfied" to "very satisfied"
Clinical results : range of mobility of the prosthetic knee | One year after surgery
  Range of motion from hyperextension to flexion (degrees)
Clinical results : complication rate | One year after surgery
  Complication rate (percentage) : manipulation under anesthesia, re-operation, revision, previous pain syndrome
Imaging results : EOS 3D, alignement of the lower limb | One year after surgery
  measurement of the frontal alignment of the lower limb (hip-knee-ankle and hip-knee-calcaneus angles)
Imaging results : EOS 3D, orientation of the implants | One year after surgery
  - measurement of the orientation of the implants in the frontal (medial proximal tibial, lateral distal femoral and joint line convergence angles) and sagittal (tibial slope, flexion of the femoral component) planes
Imaging results : EOS 3D, distance between anterior femoral cortex and prosthetic trochlea | One year after surgery
  measurement of the distance between the anterior femoral cortex and the prosthetic trochlea
Imaging results : radiography, evaluation of implant fixation | One year after surgery
  evaluation of implant fixation (e.g. sealing, border, reactive line)
Imaging results : radiography, measurement of patellar height | One year after surgery
  measurement of patellar height (pre- and post-op Caton-Deschamps index comparison)
Imaging results : radiography, evaluation of the bone structure | One year after surgery
  evaluation of bone structure (e.g. osteolysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport Bordeaux Merignac, Mérignac, France

IPD SHARING:
Plan to Share IPD: No